CLINICAL TRIAL: NCT02034864
Title: Comparison of the Effectiveness of 2 Manual Therapies on Functional Outcome in Sub-acute and Chronic Non-specific Low Back Pain at 3 Months : a Randomised Controlled Trial
Brief Title: Comparison of the Effectiveness of 2 Manual Therapies on Functional Outcome in Sub-acute and Chronic Non-specific Low Back Pain
Acronym: LC OSTEO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government); Université Paris Cité (Other); University of Paris 5 - Rene Descartes (Other); Institut Universitaire Romand de Sante au Travail (Other); URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P110142
Record Dates: First submitted 2014-01-10; First posted 2014-01-14 (Estimated); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Subacute and Chronic Non-specific Low Back Pain
Keywords: low back pain; manual therapy; randomized controlled trial
MeSH Terms: conditions — Low Back Pain | interventions — Manipulation, Osteopathic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Osteopathic manipulative treatment (Experimental): 6 sessions of standardized manipulative treatment
  Interventions: Other: Osteopathic manipulative treatment
- Placebo of osteopathic manipulative treatment (Sham Comparator): 6 sessions of standardized placebo of manipulative treatment
  Interventions: Other: Placebo of osteopathic manipulative treatment

INTERVENTIONS:
Other: Osteopathic manipulative treatment — A standardized manipulative treatment according to the results of a physical examination including 7 anatomical areas will be given by trained osteopaths during 6 sessions (with an interval of 2 weeks between 2 sessions). Each session will last 45 minutes. Osteopaths will have 3 days of training in standardized manipulative treatment.
  Arms: Osteopathic manipulative treatment
Other: Placebo of osteopathic manipulative treatment — A standardized placebo of manipulative treatment consisting in "light touch" and according to the results of a physical examination including 7 anatomical areas will be given by trained osteopaths during 6 sessions (with an interval of 2 weeks between 2 sessions). Each session will last 45 minutes. Osteopaths will have 3 days of training in standardized placebo of manipulative treatment.
  Arms: Placebo of osteopathic manipulative treatment

SUMMARY:
The purpose of this study is to determine whether a standardised osteopathic manipulative treatment is more effective than a placebo of osteopathic manipulative treatment, in sub-acute and chronic non-specific low back pain on functional recovery at 3 months.

DETAILED DESCRIPTION:
Sub-acute (4-12-week duration) and chronic (more than 3-month duration) non-specific low back pain (LBP) is frequent, disabling and costly. The effectiveness of usual treatments (including pain killers, anti-inflammatory drugs, spinal injections, physiotherapy, spinal traction, transcutaneous electrical nerve stimulation, etc) may be not sufficient, and many patients resort to alternative therapies. Manipulative treatments represent en emerging therapy in this area, although studies assessing their effectiveness are limited and often biased. The purpose of this study is to evaluate the efficacy of two manual therapies on improving functional recovery in sub-acute and chronic non-specific low back pain at 3 months. A standardised osteopathic manipulative treatment is compare to a placebo of osteopathic manipulative treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patient consulting for subacute and chronic non-specific low
* Male or female aged from 18 to 65 years (included)
* Patient can speak and understand French
* Patient giving his informed consent to participate in the study
* Patient affiliated to or beneficiary of social insurance

Exclusion Criteria:

* Specific low-back pain caused by inflammatory, tumoral, infectious disease or a back traumatism in the 3 past months
* History of back surgery and/or vertebral fracture in the previous 6 months
* Presence of a motor impairment related to the reason for consultation
* The patient is a student or a practitioner in manipulative therapies
* Pregnancy
* Inability to understand the process of the study
* The patient is already included in another clinical study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2014-02-17 (Actual); Primary Completion 2017-10-23 (Actual); Study Completion 2017-10-23 (Actual)

PRIMARY OUTCOMES:
Mean improvement from baseline in mean activity limitation | 3 months after randomization
  Assessed with the self-administered Quebec functional scale (from 0, no limitation to 100, maximal limitation)

SECONDARY OUTCOMES:
Mean reduction from baseline in mean lumbar pain in the previous 48 hrs | 3 months after randomization
  assessed with a self-administered 11-class numeric scale (from 0 no pain to 100, maximal pain)
Mean reduction from baseline in mean lumbar pain in the previous 48 hrs | 12 months after randomization
  assessed with a self-administered 11-class numeric scale (from 0, no pain to 100, maximal pain)
Number of sick leaves | 12 months after randomization
  self-reported number of sick leaves
Duration of sick leaves | 12 months after randomization
  self-reported total duration (days) of sick leaves
Recurrence of pain | 12 months after randomization
  self-reported number of low back pain episodes
Mean improvement from baseline in mean activity limitation | 12 months after randomization
  Assessed with the self-administered Quebec functional scale (from 0, no limitation to 100, maximal limitation)
Mean improvement from baseline in mean quality of life | 3 months after randomization
  Assessed with the physical and mental components of the self-administered MOS SF-12 questionnaire (from 0, worse quality of life to 100, best quality of life)
Mean improvement from baseline in mean quality of life | 12 months after randomization
  Assessed with the physical and mental components of the self-administered MOS SF-12 questionnaire (from 0, worse quality of life to 100, best quality of life)
Pain killer and non-steroidal anti-inflammatory drug consumption | 3 months after randomization
  self-reported consumption of pain killer and non-steroidal anti-inflammatory drugs since last contact ( yes/no)
Pain killer and non-steroidal anti-inflammatory drug consumption | 12 months after randomization
  self-reported consumption of pain killer and non-steroidal anti-inflammatory drugs since last contact ( yes/no)

CONTACTS AND LOCATIONS:
Overall Officials: Francois Rannou, MD PhD, Principal Investigator — AP-HP, Descartes University, INSERM
Locations (1):
- CHU Cochin, Paris, France

REFERENCES:
- [Background] Nguyen C, Boutron I, Zegarra-Parodi R, Baron G, Alami S, Sanchez K, Daste C, Boisson M, Fabre L, Krief P, Krief G, Lefevre-Colau MM, Rannou F. Effect of Osteopathic Manipulative Treatment vs Sham Treatment on Activity Limitations in Patients With Nonspecific Subacute and Chronic Low Back Pain: A Randomized Clinical Trial. JAMA Intern Med. 2021 May 1;181(5):620-630. doi: 10.1001/jamainternmed.2021.0005. PMID 33720272
- [Background] 1. Poiraudeau S, Lefèvre-Colau M.-M, Fayad F., Rannou F, Revel M. Lombalgie. Encyclopédie Médico-Chirurgicale 15-840-C-10 (2004)
- [Background] Chou R, Huffman LH; American Pain Society; American College of Physicians. Medications for acute and chronic low back pain: a review of the evidence for an American Pain Society/American College of Physicians clinical practice guideline. Ann Intern Med. 2007 Oct 2;147(7):505-14. doi: 10.7326/0003-4819-147-7-200710020-00008. PMID 17909211
- [Background] Nelemans PJ, de Bie RA, de Vet HC, Sturmans F. WITHDRAWN: Injection therapy for subacute and chronic benign low-back pain. Cochrane Database Syst Rev. 2007 Jul 18;(2):CD001824. doi: 10.1002/14651858.CD001824.pub2. PMID 17636686
- [Background] Hayden JA, van Tulder MW, Malmivaara AV, Koes BW. Meta-analysis: exercise therapy for nonspecific low back pain. Ann Intern Med. 2005 May 3;142(9):765-75. doi: 10.7326/0003-4819-142-9-200505030-00013. PMID 15867409
- [Background] Costa LO, Maher CG, Latimer J, Hodges PW, Herbert RD, Refshauge KM, McAuley JH, Jennings MD. Motor control exercise for chronic low back pain: a randomized placebo-controlled trial. Phys Ther. 2009 Dec;89(12):1275-86. doi: 10.2522/ptj.20090218. Epub 2009 Nov 5. PMID 19892856
- [Background] Lambeek LC, van Mechelen W, Knol DL, Loisel P, Anema JR. Randomised controlled trial of integrated care to reduce disability from chronic low back pain in working and private life. BMJ. 2010 Mar 16;340:c1035. doi: 10.1136/bmj.c1035. PMID 20234040
- [Background] Lindell O, Johansson SE, Strender LE. Subacute and chronic, non-specific back and neck pain: cognitive-behavioural rehabilitation versus primary care. A randomized controlled trial. BMC Musculoskelet Disord. 2008 Dec 30;9:172. doi: 10.1186/1471-2474-9-172. PMID 19116007
- [Background] Macario A, Pergolizzi JV. Systematic literature review of spinal decompression via motorized traction for chronic discogenic low back pain. Pain Pract. 2006 Sep;6(3):171-8. doi: 10.1111/j.1533-2500.2006.00082.x. PMID 17147594
- [Background] Assendelft WJ, Morton SC, Yu EI, Suttorp MJ, Shekelle PG. Spinal manipulative therapy for low back pain. A meta-analysis of effectiveness relative to other therapies. Ann Intern Med. 2003 Jun 3;138(11):871-81. doi: 10.7326/0003-4819-138-11-200306030-00008. PMID 12779297
- [Background] Bronfort G, Haas M, Evans RL, Bouter LM. Efficacy of spinal manipulation and mobilization for low back pain and neck pain: a systematic review and best evidence synthesis. Spine J. 2004 May-Jun;4(3):335-56. doi: 10.1016/j.spinee.2003.06.002. PMID 15125860
- [Background] Manheimer E, White A, Berman B, Forys K, Ernst E. Meta-analysis: acupuncture for low back pain. Ann Intern Med. 2005 Apr 19;142(8):651-63. doi: 10.7326/0003-4819-142-8-200504190-00014. PMID 15838072
- [Background] Rubinstein SM, van Middelkoop M, Kuijpers T, Ostelo R, Verhagen AP, de Boer MR, Koes BW, van Tulder MW. A systematic review on the effectiveness of complementary and alternative medicine for chronic non-specific low-back pain. Eur Spine J. 2010 Aug;19(8):1213-28. doi: 10.1007/s00586-010-1356-3. Epub 2010 Mar 14. PMID 20229280
- [Background] Licciardone JC, Brimhall AK, King LN. Osteopathic manipulative treatment for low back pain: a systematic review and meta-analysis of randomized controlled trials. BMC Musculoskelet Disord. 2005 Aug 4;6:43. doi: 10.1186/1471-2474-6-43. PMID 16080794
- [Background] Andersson GB, Lucente T, Davis AM, Kappler RE, Lipton JA, Leurgans S. A comparison of osteopathic spinal manipulation with standard care for patients with low back pain. N Engl J Med. 1999 Nov 4;341(19):1426-31. doi: 10.1056/NEJM199911043411903. PMID 10547405
- [Background] Licciardone JC, Stoll ST, Fulda KG, Russo DP, Siu J, Winn W, Swift J Jr. Osteopathic manipulative treatment for chronic low back pain: a randomized controlled trial. Spine (Phila Pa 1976). 2003 Jul 1;28(13):1355-62. doi: 10.1097/01.BRS.0000067110.61471.7D. PMID 12838090
- [Background] Hoehler FK, Tobis JS, Buerger AA. Spinal manipulation for low back pain. JAMA. 1981 May 8;245(18):1835-8. PMID 6453240
- [Background] Schulz KF, Altman DG, Moher D; CONSORT Group. CONSORT 2010 statement: updated guidelines for reporting parallel group randomised trials. BMJ. 2010 Mar 23;340:c332. doi: 10.1136/bmj.c332. PMID 20332509
- [Background] Boutron I, Moher D, Altman DG, Schulz KF, Ravaud P; CONSORT Group. Extending the CONSORT statement to randomized trials of nonpharmacologic treatment: explanation and elaboration. Ann Intern Med. 2008 Feb 19;148(4):295-309. doi: 10.7326/0003-4819-148-4-200802190-00008. PMID 18283207
- See also: World Health Organization Benchmarks for training in osteopathy. Novembre 2010. Site Internet de l'Organisation Mondiale de la Santé — http://whqlibdoc.who.int/publications/2010/9789241599665_eng.pdf
- See also: Official Journal of the European Union Website. Directive 2005/36/EC of the European Parliament and of the Council of 7 September 2005 on the recognition of professional qualifications p. 22-142 — http://eur-lex.europa.eu/LexUriServ/LexUriServ.do?uri=OJ:L:2005:255:0022:0142:en:PDF